CLINICAL TRIAL: NCT01814618
Title: Trial of Directed High-dose Nasal Steroids on Residual Olfactory Dysfunction in Patients With Chronic Rhinosinusitis Following Endoscopic Sinus Surgery
Brief Title: Trial of Directed High-dose Nasal Steroids on Residual Smell Loss in Sinus Patients After Sinus Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1567
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2014-09

CONDITIONS: Olfaction Disorders; Sinusitis; Paranasal Sinus Diseases
MeSH Terms: conditions — Olfaction Disorders; Sinusitis; Paranasal Sinus Diseases | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): These subjects did not have improved sense of smell after surgery and were randomized to this observation group or treatment group. These patients will be observed post-operatively but will not receive the trial medication.
- Treatment (Experimental): These subjects did not have improved sense of smell after surgery and were randomized to this treatment group or the observation. These patients will be observed post-operatively and will receive a 3-month course of topical nasal steroids(budesonide respules).
  Drug: Budesonide Respules
  Other Names:
  Pulmicort respules
  Subjects irrigate their noses with budesonide respules. They will use one respule per nostril twice daily for three months.
  Interventions: Drug: Budesonide Respules

INTERVENTIONS:
Drug: Budesonide Respules — Subjects irrigate their noses with budesonide respules. They will use one respule per nostril twice daily for three months.
  Other Names: Pulmicort respules
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine if a trial of directed high-dose nasal steroids improves residual smell loss in patients with chronic rhinosinusitis following sinus surgery. Other outcomes of this study include: identifying the differences in sinus airflow between patients who improve following nasal steroid treatment and those who do not, and to see if, in patients who improve following surgery, the improvement remains throughout follow-up.

DETAILED DESCRIPTION:
OVERVIEW:

This is a prospective randomized cohort study assessing the use of directed high-dose nasal steroids for improving olfactory function after endoscopic sinus surgery for chronic rhinosinusitis. Up to 70 subjects will be prospectively enrolled from patients visiting the Department of Otolaryngology-Head and Neck Surgery clinics at the University of North Carolina (UNC) Hospitals.

VISIT 1/PRE-OPERATIVE VISIT

Visit 1 will be the day of enrollment or the pre-operative visit. During this encounter, subjects will complete the Rhinosinusitis Disability Index (RSDI), Rhinosinusitis Outcome Measure 31 (RSOM-31), Sinonasal Outcome Test 22 (SNOT-22), University of Pennsylvania Smell Identification Test (UPSIT), Phenyl-ethyl-alcohol (PEA) tests and will also have their Lund-Kennedy scores recorded. Additionally, all subjects will undergo a pre-operative (standard of care) head CT which will be scored with the Lund-Mackay system. This standard of care head CT will be billed to the subject's insurance.

VISIT 2/POST-OPERATIVE VISIT(POV) 1

Visit 2 will occur at "post-operative visit 1" or 4-6 weeks after surgery. During this encounter, subjects will complete the RSDI, RSOM-31, SNOT-22, UPSIT, PEA tests and will also have their Lund-Kennedy scores recorded. Additionally, all subjects will undergo post-operative (standard of care) head CT. This standard of care head CT will be billed to the subject's insurance. Subjects who do have quantitative improvement in olfaction (as determined by UPSIT category score) will be considered part of the "improved" group and will simply be followed without an intervention. Subjects who do not have quantitative improvement in olfaction will be randomized (with a random number generator) into a "treatment" or an "observation" group. Subjects within the treatment group will be given a 12-week course of directed high-dose nasal steroid irrigation. Pharmacies will bill the subjects' insurance for the medication. Subjects will be instructed to perform irrigation twice daily using ½ budesonide respule, 0.5 mg/2mL, applied directly to the nasal mucosa as described previously. Subjects will be given written instructions on how to perform nasal irrigation with this medication. Subjects randomized to receive medication will be given medication diaries and asked to document medication compliance and side effects.

PHONE INTERVIEW (1-2 WEEKS AFTER TREATMENT)

Subjects randomized to the treatment arm will be called 1-2 weeks after initiation of budesonide treatment to assess medication compliance and side effects. Subjects will be asked to review their medication diaries when answering questions about compliance and side effects. As detailed in the data safety monitoring plan, the PI will be alerted if any subjects are experiencing moderate-severe adverse events or any unexpected side effects.

VISIT 3/"SURVEILLANCE" VISIT

Visit 3 will be a surveillance visit somewhere between post-operative visit 1 (at 4-6 weeks) and post-operative visit 2 (at 3-4 months). Only patients in the treatment arm will have this visit. During this visit, subjects will be asked about medication compliance and asked to demonstrate irrigation technique with nasal saline. Medication diaries will be reviewed and assessed for compliance and concerning side effects. These diaries will be collected for future review by the independent data safety reviewer.

VISIT 4/ POST-OPERATIVE VISIT (POV) 2

Visit 4 will occur at post-operative visit 2 or 3-4 months after surgery. During this encounter, subjects will complete the RSDI, RSOM-31, SNOT-22, UPSIT, PEA tests and will also have their Lund-Kennedy scores recorded. Subjects in the "non-improved" arm (regardless of whether they were randomized to receive nasal steroids) will have an additional (for research purposes only) head CT. This research only head CT will be provided free of charge by the Department of Otolaryngology's CT scanner.

Medication diaries will be reviewed and assessed for compliance and concerning side effects. These diaries will be collected for future review by the independent data safety reviewer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are otherwise healthy undergoing surgery for treatment of chronic rhinosinusitis will be evaluated for olfactory dysfunction, and if present, will be recruited for study participation. The subjects will be included without regard to their gender, race or ethnicity. Subjects will be identified from patients in the clinical practices of the Department of Otolaryngology - Head and Neck Surgery at the University of North Carolina. Only adult patients greater than 18 years old and less than 85 will be approached for this study, as patient treatment algorithms outside this range tend to vary with greater frequency. Due to limited resources, only patients fluent in English will be included, thus minimizing confounding variables and hurdles to patient communication, as some clinics do not have interpreting services. Also, most of the quality of life surveys and olfactory testing do not have non English versions. Only patients with health insurance will be included in the study in order to ensure all participants have access to the study drug.

Exclusion Criteria:

* If the patient is a premenopausal woman, she will be asked if she is pregnant or breastfeeding. If she is either of these, she will be excluded from the study. All remaining women will receive a urine pregnancy test. If this urine pregnancy test is positive, the patient will be excluded from the study. Thus, for premenopausal female patients, a negative urine pregnancy test is necessary for inclusion in the study because of the need for repeat CTs and the possible systemic manifestations due to steroid irrigation. Further exclusion criteria will include the following: hypersensitivity to cortisol, history of pituitary disease, and allergic disease with subsequent anaphylaxis or breathing difficulties. Additionally, patients with a history of immunodeficiency, autoimmune disease, cystic fibrosis, or previous sinus surgery will be excluded as these co-morbidities might cloud the relationship between the treatment and the outcome.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Degree of Olfactory Function | 4-6 week post-operative visit
  Measurements of smell will be taken at the initial preoperative visit and again at the 4-6 week postoperative visit using the University of Pennsylvania Smell Identification Test (UPSIT) and the Phenyl Ethyl Alcohol (PEA) Threshold test, in which smell is assessed by smelling different concentrations of PEA. The UPSIT is a scratch and sniff test and the PEA threshold testing is a process by which the subject smells vials of different concentrations of odorant (PEA) to determine lowest detectable concentration of odorant.
Change in Degree of Olfactory Function | 3-4 month post-operative visit
  Measurements of smell will be taken at the initial preoperative visit and again at the 3-4 month postoperative visit using the University of Pennsylvania Smell Identification Test (UPSIT) and the Phenyl Ethyl Alcohol (PEA) Threshold test, in which smell is assessed by smelling different concentrations of PEA. The UPSIT is a scratch and sniff test and the PEA threshold testing is a process by which the subject smells vials of different concentrations of odorant (PEA) to determine lowest detectable concentration of odorant.

SECONDARY OUTCOMES:
Change in Head CT Grade | 4-6 week post-operative visit
  A head CT will be performed at the initial preoperative visit and at the 4-6 week post-operative visit. The head CT will be assessed using the Lund-Mackay scoring system, in which physician graders will analyze the CT for abnormalities in the patient's sinuses and nasal cavity.
Change in Head CT Grade | 3-4 month post-operative visit
  Subjects in the "non-improved" arm (regardless of whether they were randomized to receive nasal steroids) will receive a head CT at this time point. The CT will be assessed using the Lund-Mackay scoring system, in which physician graders will analyze the CT for abnormalities in the patient's sinuses and nasal cavity.
Change in Nasal Endoscopy Grade | 4-6 week post-operative visit
  Nasal endoscopy will be performed at the initial preoperative visit and again at the 4-6 week postoperative visit. The nasal cavity and sinuses will be assessed using the Lund-Kennedy scoring method which addresses crusting, scarring, edema, discharge, and presence of polyps.
Change in Nasal Endoscopy Grade | 3-4 month post-operative visit
  Nasal endoscopy will be performed at the initial preoperative visit and at the 3-4 month postoperative visit. The nasal cavity and sinuses will be assessed using the Lund-Kennedy scoring method which addresses crusting, scarring, edema, discharge, and presence of polyps.
Change in Quality of Life | 4-6 week post-operative visit
  Quality of life will be assessed at the initial preoperative visit as well as the 4-6 week postoperative visit using the Sinonasal Outcome Test 22(SNOT-22) and the Rhinosinusitis Outcome Measure 31 (RSOM-31). The Snot-22 and RSOM-31 are questionnaires used to measure disease related quality of life and symptoms.
Change in Quality of Life | 3-4 month post-operative visit
  Quality of life will be assessed at the initial preoperative visit as well as the 3-4 month postoperative visit using the Sinonasal Outcome Test 22(SNOT-22) and the Rhinosinusitis Outcome Measure 31 (RSOM-31). The Snot-22 and RSOM-31 are questionnaires used to measure disease related quality of life and symptoms.
Number of patients with steroid side effects after a 1-2 week course of steroids | 5-8 weeks post-operatively
  Subjects who were randomized to the treatment arm will be contacted by phone 1-2 weeks after starting steroids and will review a pre-constructed medication safety and side effect questionnaire with the caller. Patients will also be asked to review their medication diary with the caller.
Number of patients with steroid side effects after a 8 week course of steroids | 3-4 month post-operative visit
  Subjects who were randomized to the treatment arm will return to clinic 3-4 months postoperatively and medication diaries will be reviewed and assessed for compliance and concerning side effects. These diaries will be collected for future review by the independent data safety reviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Zanation, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill Department of Otolaryngology/Head and Neck Surgery, Chapel Hill, North Carolina, United States